CLINICAL TRIAL: NCT04713748
Title: Pilot Study to Compare Serology Results From Blood Collected Using Tasso-SST OnDemand Device Compared to Venipuncture
Brief Title: Tasso-SST OnDemand Comparator Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00107313
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Results first posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: C3PI Study Testing Group
Keywords: Tasso-SST

STUDY DESIGN:
Intervention Model Description: Participants will collect a small blood sample using the Tasso-SST OnDemand device during a serology blood draw visit already scheduled for the MURDOCK C3PI Study (Pro00105703). Participants will be provided a kit that includes written, step-by-step instructions that include pictures. Participants will also have the option to watch a brief video on using the device, available online, prior to collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Tasso- SST blood collection (Other): About 100 participants will have blood collected by two methods-regular phlebotomy and Tasso-SST, in this pilot study.
  Interventions: Device: Tasso-SST on Demand
- Regular Venipuncture (Other): About 100 participants will have blood collected by two methods-regular phlebotomy and Tasso-SST, in this pilot study.
  Interventions: Other: Regular Phlebotomy

INTERVENTIONS:
Device: Tasso-SST on Demand — Participants will collect a small blood sample using the Tasso-SST OnDemand device during a serology blood draw visit already scheduled for the MURDOCK C3PI Study (Pro00105703). Participants will be provided a kit that includes written, step-by-step instructions that include pictures. Participants will also have the option to watch a brief video on using the device, available online, prior to collection. Both blood samples will be spun and processed for serum. Serum will be frozen and shipped to the lab at Duke for antibody testing. Antibody results will be compared between the two methods.
  Arms: Tasso- SST blood collection
Other: Regular Phlebotomy — Participants will have a small blood sample collected via regular venipuncture.
  Arms: Regular Venipuncture

SUMMARY:
Purpose and objective: The purpose of this pilot study is participant user acceptance testing of the Tasso-SST OnDemand device to collect blood for antibody testing. The study will also compare antibody testing results from blood collected using the Tasso-SST OnDemand device compared to blood collected by phlebotomy.

Study activities and population group: All participants enrolled in the MURDOCK C3PI Study (Pro Pro00105703), and actively participating in the testing cohort (n=300), will be emailed about the study. One or more reminder emails may be sent. The study seeks to enroll up to 100 participants.

Participants will collect blood using the Tasso-SST OnDemand at the same visit where blood will be collected via phlebotomy for the MURDOCK C3PI study. Blood samples will be spun and processed for serum, which will be shipped frozen to analytical lab at Duke. Participants will complete a short survey about their experience using the Tasso-SST OnDemand device.

Data analysis and risk/safety issues: The study team will evaluate correlation between results from blood collected by the two methods and qualitatively exam participant survey results. There are no risk/safety issues. Risk of reaction at the collection site is similar to that of phlebotomy and is described in the electronic consent form.

DETAILED DESCRIPTION:
Purpose: The purpose of this pilot study is participant user acceptance testing of the Tasso-SST OnDemand device to collect blood for antibody testing. The study will also compare antibody testing results from blood collected using the Tasso-SST On-Demand device compared to blood collected by phlebotomy.

Design and Procedure: Participants will collect a small blood sample using the Tasso-SST OnDemand device during a serology blood draw visit already scheduled for the MURDOCK C3PI Study (Pro00105703). Participants will be provided a kit that includes written, step-by-step instructions that include pictures. Participants will also have the option to watch a brief video on using the device, available online, prior to collection. The Tasso-SST OnDemand device collects whole capillary blood, at a minimum volume of 80ul.

A standard blood draw will also be done and both blood samples will be spun and processed for serum. Serum will be frozen and shipped to the lab at Duke for antibody testing. Antibody results will be compared between the two methods.

Participants will be sent a brief survey to learn about their experience using the Tasso-SST OnDemand device.

Selection of Subject:

Subject Recruitment: All participants meeting eligibility criteria will be emailed about the study. One or more reminder emails may be sent about the study. The study seeks to enroll up to 100 participants.

The Tasso-SST OnDemand device sticks to the skin with a light adhesive. When the button is pressed, a vacuum forms and a lancet pricks the surface of the skin. The vacuum draws blood out of the capillaries and into a tube attached to the bottom of the device. The Investigator Brochure is attached to this submission.

Risk and Benefit Assessment: The Tasso-SST OnDemand device uses an adhesive - the device should be removed immediately if there are any signs of an allergic reaction. There is risk of bruising or soreness at the site where blood is drawn. There is also a slight possibility of infection, and a rare risk of fainting.

Participants can minimize risk by closely following the instructions provided with the kits.

Trained staff will be present should the participant have any concerns or issues.

The study does not have a direct benefit to participants. The information learned could lead to future use of the Tasso-SST OnDemand device to collect blood safely at home.

Data Analysis and Data Safety Monitoring: The study team will evaluate correlation between results from blood collected by the two methods in this pilot study and qualitatively exam participant survey results. Summary statistics will be generated for survey responses, and qualitative data will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Must be a study participant enrolled in the MURDOCK C3PI Study (Pro00105703), participating in the testing cohort of the study.
* Participants are therefore 18 years of age or older, and
* willing to read and complete the consent process.

Exclusion Criteria:

* No exclusion criteria; however, only up to 100 participants will be enrolled. If more than 100 participants sign consent, some interested participants may not take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L.Kristin Newby, MD, MHS, Principal Investigator — Duke University
Locations (1):
- Duke CTSI Translational Population Health Office, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. Recruitment into the Tasso Pilot Study occurred from 1/15/2021 to 3/10/2021.
  2. All participants were recruited from tC3PI Study sub-cohort - had serial COVID-19 bimonthly antibody testing.
  3. A total of 281 participants in the C3PI invited to participate.
  4. 135 eligible individuals provided consent for the Tasso Pilot Study.
Groups:
- TASSO-SST OnDemand Blood Collection vs. Routine Phlebotomy: Compared the performance of TASSO-SST OnDemand blood collection with routine phlebotomy (gold standard) on paired samples from the same participant.
Period: Overall Study
Arm/Group | TASSO-SST OnDemand Blood Collection vs. Routine Phlebotomy
Started | 135
Completed | 100
Not Completed | 35
Not completed — Not enough kits allocated | 35

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | TASSO-SST OnDemand Blood Collection vs. Routine Phlebotomy
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 67
  >=65 years | 33
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.5 [47.5 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 93
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 85
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity is Calculated as the Percentage of the Abbott Alinity Nucleocapsid IgG Antibody Assay Positive Cases Testing Positive Using TASSO-SST Collected Blood Samples. Se=N Tasso(+) / N Phlebotomy Antibody (+) Assay (+)
Description: Sensitivity is defined as the number detected as positive on the new screen (Tasso) divided by the number defined as positive under the 'gold standard' multiplied by 100%. This is presented as a comparison to testing of blood samples obtained by routine phlebotomy as the gold standard (Abbott Alinity nucleocapsid IgG antibody assay drawn by a phlebotomist).
Time Frame: up to 17 days after onset of symptoms
Population: Participants who were able to draw blood using the TASSO-SST OnDemand device.
Measure: Number; unit: percent sensitivity
Arm/Group | TASSO-SST OnDemand Blood Collection vs. Routine Phlebotomy
Number analyzed (Participants) | 70
percent sensitivity | 100

2. Primary Outcome: Reliability of the Abbott Alinity Nucleocapsid IgG Antibody Assay Using TASSO-SST Collected Blood Samples
Description: Interclass correlation (ICC) uses the 2 measures (Tasso & SST), measured on the same subjects. ICC is defined as the Variance between Persons (Var-P) divided by the Variance within Persons (error) Var-E.
  ICC is defined as Var-P/(Var-P + Var-E). confidence intervals are easily defined by incorporating sample size.
  Presented as the interclass correlation coefficient between TASSO-SST collected and routine phlebotomy sample results.
Time Frame: up to 17 days after onset of symptoms
Population: Participants who were able to draw blood using the TASSO-SST OnDemand device.
Measure: Number (95% Confidence Interval); unit: interclass correlation coefficient
Arm/Group | TASSO-SST OnDemand Blood Collection vs. Routine Phlebotomy
Number analyzed (Participants) | 70
interclass correlation coefficient | 0.98 [0.97 to 0.99]
Statistical Analysis 1: Comparison: TASSO-SST OnDemand Blood Collection vs. Routine Phlebotomy; Test type: Other; p < 0.0001, Interclass correlation coefficient

3. Primary Outcome: Bias Between TASSO-SST Collected Blood Samples and Routine Phlebotomy Samples in the Abbott Alinity Nucleocapsid IgG Antibody Assay
Description: Bias is measured using the Bland-Altman method. Here, the difference the values by the 2 measures (Phlebotomy-Tasso) (difference) is compared to the average of Phlebotomy & Tasso (average). Bias is defined as differences which vary from 0, and is measured by (1) assessing if the average difference is non-zero, and (2) if the difference is systematically more or less close to 0 as the average increases. Presented as the regression slope.
Time Frame: up to 17 days after onset of symptoms
Population: Participants who were able to draw blood using the TASSO-SST OnDemand device.
Measure: Mean (Standard Deviation); unit: slope
Arm/Group | TASSO-SST OnDemand Blood Collection vs. Routine Phlebotomy
Number analyzed (Participants) | 70
slope | 0.72 (1.42)

ADVERSE EVENTS:
Time Frame: 1 day per patient.
Groups:
- Definition of Arm/Group: This is a single armed trial comparing 2 measures for COVID determination in a clinical sample.
Arm/Group | Definition of Arm/Group
All-Cause Mortality (participants affected / at risk) | 0/135
Serious Adverse Events (participants affected / at risk) | 0/135
Other Adverse Events (participants affected / at risk) | 0/135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT04713748/Prot_SAP_000.pdf